CLINICAL TRIAL: NCT03846453
Title: A Phase 3, Multicenter, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of 0.25% HL036 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye
Brief Title: A Study to Assess Efficacy and Safety of HL036 in Subjects With Dry Eyes
Acronym: VELOS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL036-DED-US-P301
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.25% HL036 Ophthalmic Solution (Experimental): Participants self-administered HL036 0.25% ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment (CAE®) were conducted at Day 1, Day 15, Day 29 and Day 57
  Interventions: Biological: HL036 Ophthalmic Solution
- Placebo (Placebo Comparator): Participants self-administered HL036 placebo (vehicle solution) as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HL036 Ophthalmic Solution — HL036 Ophthalmic Solution
  Other Names: Tanfanercept
  Arms: 0.25% HL036 Ophthalmic Solution
Biological: Placebo — Placebo vehicle solution
  Arms: Placebo

SUMMARY:
The objective of this study was to compare the safety and efficacy of 0.25% HL036 Ophthalmic Solutions to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have a patient-reported history of dry eye for at least 6 months prior to Visit 1
* Be willing and able to comply with all study procedures
* Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2

Exclusion Criteria:

* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months
* Have any previous experience using HL036

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Eye Research Foundation, Newport Beach, California
  - East West Eye Institute, Torrance, California
  - Specialty Retina Center, Boynton Beach, Florida
  - Specialty Retina Center, Coral Springs, Florida
  - Eye Care Centers Management Inc, Morrow, Georgia
  - MidWest Cornea Associates, LLC, Indianapolis, Indiana
  - The Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Vita Eye Clinic, Shelby, North Carolina
  - Total Eye Care, P A, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the eligibility criteria were enrolled at 12 sites in the United States.
Pre-assignment Details: A total of 1108 patients were screened and 637 patients were enrolled and randomized to one of the treatment groups. The enrollment number in Protocol refers to the participants randomized to the treatment group.
Groups:
- Placebo-Run in Participants: All participants entered placebo-run in period for 14 days prior to randomization. During the period, exposures to the CAE were conducted to ascertain eligibility to enter the study. Those who qualified were randomized to either 0.25% HL036 Ophthalmic Solution group or placebo group.
- 0.25% HL036 Ophthalmic Solution: Participants self-administered HL036 0.25 % ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment (CAE®) were conducted at Day 1, Day 15, Day 29 and Day 57.
Period: Placebo Run-in (14 Days)
Arm/Group | Placebo-Run in Participants | 0.25% HL036 Ophthalmic Solution | Placebo
Started | 1108 | 0 (Participants in this group were randomized after they completed the placebo run-in period.) | 0 (Participants in this group were randomized after they completed the placebo run-in period.)
Completed | 637 | 0 | 0
Not Completed | 471 | 0 | 0
Not completed — Eligibility Criteria Not Met | 465 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Other | 2 | 0 | 0
Period: Randomized Treatment Period (Days 57±3)
Arm/Group | Placebo-Run in Participants | 0.25% HL036 Ophthalmic Solution | Placebo
Started | 0 (All participants who completed the placebo run-in period and qualified were randomized to either 0.25% HL036 Ophthalmic Solution group or placebo group.) | 318 | 319
Completed | 0 | 291 | 294
Not Completed | 0 | 27 | 25
Not completed — Adverse Event | 0 | 16 | 8
Not completed — Protocol Violation | 0 | 6 | 5
Not completed — Administrative Reasons | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 4
Not completed — Other | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: The intent-to-treat (ITT) population includes all randomized participants.
Groups:
- 0.25% HL036 Ophthalmic Solution: Participants self-administered HL036 0.25 percent (%) ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 1, Day 15, Day 29 and Day 57.
- Placebo: Participants sefl-administered HL036 placebo matching vehicle solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 1, Day 15, Day 29 and Day 57.
- Total: Total of all reporting groups
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 318 | 319 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.86) | 62.9 (14.02) | 62.0 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 211 | 441
  Male | 88 | 108 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 25 | 49
  Not Hispanic or Latino | 294 | 294 | 588
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 18 | 19 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 53 | 124
  White | 228 | 238 | 466
  More than one race | 1 | 7 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Coprimary Endpoint: Change From Baseline in Inferior Corneal Fluorescein Staining Score to Day 57 (Pre- to Post-CAE)
Description: It was evaluated for the inferior region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: Pre-CAE and Post-CAE on Day 1 (Baseline) and Day 57
Population: ITT Population with the Markov Chain Monte Carlo (MCMC) imputation method for missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.38 (0.427) | 1.31 (0.411)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.47 (0.900) | -0.52 (0.762)
Statistical Analysis 1: Comparison: 0.25% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.1871, ANCOVA — P-value calculated using a model with treatment, baseline score, and site as covariates; Least Squares (LS) Mean Difference = 0.08, 95% CI 2-sided [-0.04 to 0.21], Standard Error of Mean 0.064

2. Primary Outcome: Coprimary Endpoint: Change From Baseline in Ocular Discomfort Score to Day 57 (Pre-CAE)
Description: It is assessed by the Ora Calibra® Ocular Discomfort scale. The score ranged from 0 to 4 (0=none and 4=severe) with 1 point increments, where lower scores indicate improvement.
Time Frame: Baseline (Day 1 Pre-CAE), Day 57 (Pre-CAE)
Population: ITT Population with the MCMC imputation method for missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 2.61 (0.975) | 2.53 (1.060)
  Change from Baseline: Day 57 (Pre-CAE) | -0.47 (1.318) | -0.47 (1.287)
Statistical Analysis 1: Comparison: 0.25% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.5549, ANCOVA; P-value calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = 0.05, 95% CI 2-sided [-0.12 to 0.23], Standard Error of Mean 0.090

3. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Inferior Region)
Description: It is evaluated for the inferior region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: Baseline (Day 1 Pre-CAE and Post-CAE), Day 8, Day 15 (Pre-CAE and Post-CAE), Day 29 (Pre-CAE and Post-CAE), and Day 57 (Pre-CAE and Post-CAE)
Population: Number of participants analyzed included participants in ITT Population with available data. The analysis was carried out with observed data only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 0.25% HL036 Ophthalmic Solution: Participants self-administered HL036 0.25 % ophthalmic solution as topical ophthalmic drops BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.78 (0.550) | 1.84 (0.527)
  Day 1 Post-CAE | 3.17 (0.548) | 3.15 (0.546)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.38 (0.427) | 1.31 (0.411)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | 0.08 (0.626) | -0.02 (0.637)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.08 (0.730) | -0.14 (0.648)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.54 (0.797) | -0.58 (0.703)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.46 (0.843) | -0.44 (0.746)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.14 (0.651) | -0.19 (0.741)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.60 (0.851) | -0.69 (0.771)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.48 (0.840) | -0.49 (0.795)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.13 (0.734) | -0.12 (0.713)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.60 (0.855) | -0.65 (0.734)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.47 (0.829) | -0.53 (0.709)

4. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Superior Region)
Description: It is evaluated for the superior region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.81 (0.617) | 1.82 (0.556)
  Day 1 Post-CAE | 2.19 (0.614) | 2.20 (0.638)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.39 (0.629) | 0.39 (0.625)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.10 (0.665) | -0.15 (0.639)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.24 (0.665) | -0.26 (0.616)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.31 (0.732) | -0.35 (0.735)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.08 (0.800) | -0.09 (0.836)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.35 (0.652) | -0.36 (0.677)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.44 (0.774) | -0.41 (0.681)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.09 (0.887) | -0.05 (0.738)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.36 (0.677) | -0.26 (0.672)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.35 (0.779) | -0.37 (0.710)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.01 (0.880) | -0.11 (0.902)

5. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Central Region)
Description: It is evaluated for the central region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.40 (0.780) | 1.36 (0.654)
  Day 1 Post-CAE | 1.63 (0.779) | 1.66 (0.721)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.22 (0.674) | 0.30 (0.552)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.14 (0.726) | -0.02 (0.746)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.24 (0.748) | -0.17 (0.694)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.23 (0.770) | -0.24 (0.742)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.00 (0.818) | -0.08 (0.757)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.38 (0.785) | -0.23 (0.737)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.38 (0.718) | -0.38 (0.643)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.01 (0.892) | -0.14 (0.753)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.32 (0.834) | -0.18 (0.758)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.25 (0.770) | -0.29 (0.687)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.07 (0.944) | -0.10 (0.867)

6. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Temporal Region)
Description: It is evaluated for the temporal region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.62 (0.701) | 1.67 (0.738)
  Day 1 Post-CAE | 1.94 (0.692) | 1.95 (0.704)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.33 (0.636) | 0.28 (0.600)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.06 (0.714) | -0.07 (0.683)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.18 (0.760) | -0.20 (0.726)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.25 (0.705) | -0.24 (0.715)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.06 (0.840) | -0.05 (0.801)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.12 (0.700) | -0.11 (0.756)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.22 (0.691) | -0.17 (0.691)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.10 (0.852) | -0.07 (0.818)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.10 (0.775) | -0.11 (0.715)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.11 (0.730) | -0.18 (0.698)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.01 (0.907) | -0.07 (0.838)

7. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Nasal Region)
Description: It is evaluated for the nasal region on the Ora Calibra® and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.71 (0.740) | 1.73 (0.756)
  Day 1 Post-CAE | 2.10 (0.760) | 2.08 (0.813)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.39 (0.666) | 0.35 (0.663)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.04 (0.665) | -0.03 (0.673)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.13 (0.748) | -0.14 (0.690)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.20 (0.820) | -0.18 (0.797)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.07 (0.861) | -0.04 (0.883)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.11 (0.714) | -0.14 (0.733)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.23 (0.779) | -0.17 (0.787)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.12 (0.896) | -0.03 (0.837)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.11 (0.743) | -0.08 (0.706)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.16 (0.837) | -0.15 (0.760)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.06 (0.891) | -0.06 (0.886)

8. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Corneal Sum)
Description: Corneal sum score is the sum of all regions of the cornea (inferior, superior and central regions). Individual region score was evaluated on the Ora Calibra® and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Corneal sum score ranges from 0 to 12. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 4.99 (1.266) | 5.01 (1.123)
  Day 1 Post-CAE | 6.99 (1.369) | 7.01 (1.359)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.99 (1.103) | 2.00 (1.065)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.16 (1.406) | -0.18 (1.475)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.56 (1.505) | -0.57 (1.436)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -1.08 (1.673) | -1.17 (1.576)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.53 (1.646) | -0.62 (1.562)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.87 (1.475) | -0.78 (1.630)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -1.42 (1.698) | -1.47 (1.519)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.57 (1.737) | -0.68 (1.644)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.82 (1.664) | -0.56 (1.645)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -1.20 (1.840) | -1.31 (1.603)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.39 (1.853) | -0.74 (1.811)

9. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Conjunctival Sum)
Description: Conjunctival sum score is the sum of all regions of the conjunctiva (temporal and nasal regions). Individual region score was evaluated on the Ora Calibra® and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Corneal sum score ranges from 0 to 8. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 3.33 (1.327) | 3.40 (1.363)
  Day 1 Post-CAE | 4.05 (1.305) | 4.03 (1.366)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.71 (1.084) | 0.63 (1.046)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.10 (1.187) | -0.10 (1.129)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.31 (1.336) | -0.34 (1.218)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.44 (1.308) | -0.42 (1.340)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.13 (1.388) | -0.08 (1.399)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.23 (1.225) | -0.25 (1.308)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.45 (1.285) | -0.34 (1.215)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.22 (1.501) | -0.10 (1.357)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.22 (1.332) | -0.19 (1.215)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.27 (1.345) | -0.33 (1.280)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.07 (1.479) | -0.12 (1.432)

10. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining Total Score (All Five Regions: Central, Superior, Inferior, Temporal, Nasal)
Description: Total score was sum of all 5 regions: central, superior, inferior, temporal, and nasal. Individual region score was evaluated on the Ora Calibra® and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 20. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 8.33 (2.209) | 8.41 (2.075)
  Day 1 Post-CAE | 11.03 (2.164) | 11.04 (2.246)
  Day 1 (Change from Pre-CAE to Post-CAE) | 2.71 (1.668) | 2.63 (1.703)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.26 (2.191) | -0.29 (2.208)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.87 (2.462) | -0.91 (2.296)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -1.53 (2.442) | -1.59 (2.440)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.66 (2.393) | -0.70 (2.403)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -1.10 (2.298) | -1.02 (2.521)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -1.87 (2.496) | -1.82 (2.288)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.79 (2.618) | -0.78 (2.423)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -1.03 (2.522) | -0.75 (2.445)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -1.48 (2.711) | -1.64 (2.423)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.46 (2.693) | -0.86 (2.739)

11. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Score (Inferior Region)
Description: It is evaluated for the inferior region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.03 (0.720) | 1.12 (0.754)
  Day 1 Post-CAE | 1.71 (1.084) | 1.72 (1.008)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.67 (0.918) | 0.60 (0.922)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | 0.03 (0.771) | -0.05 (0.799)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.08 (0.723) | -0.13 (0.796)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.14 (1.035) | -0.18 (1.045)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.05 (1.088) | -0.05 (1.207)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.09 (0.725) | -0.21 (0.812)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.15 (1.071) | -0.19 (1.041)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.07 (1.078) | 0.01 (1.169)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.11 (0.744) | -0.21 (0.793)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.20 (1.015) | -0.25 (0.953)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.09 (1.064) | -0.03 (1.142)

12. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Score (Superior Region)
Description: It is evaluated for the superior region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 0.81 (0.710) | 0.82 (0.695)
  Day 1 Post-CAE | 0.96 (0.806) | 0.98 (0.820)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.15 (0.587) | 0.17 (0.569)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.04 (0.662) | -0.07 (0.674)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.13 (0.660) | -0.13 (0.675)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.15 (0.634) | -0.13 (0.739)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.01 (0.785) | 0.01 (0.780)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.17 (0.598) | -0.18 (0.639)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.17 (0.644) | -0.16 (0.709)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.00 (0.793) | 0.03 (0.792)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.21 (0.620) | -0.18 (0.606)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.18 (0.605) | -0.22 (0.620)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.03 (0.780) | -0.03 (0.805)

13. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Score (Central Region)
Description: It is evaluated for the central region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 0.39 (0.691) | 0.39 (0.646)
  Day 1 Post-CAE | 0.55 (0.698) | 0.57 (0.731)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.15 (0.587) | 0.18 (0.559)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.02 (0.662) | -0.04 (0.625)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.11 (0.620) | -0.04 (0.663)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.08 (0.631) | -0.08 (0.698)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.02 (0.705) | -0.04 (0.788)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 306 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.11 (0.671) | -0.08 (0.586)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.12 (0.554) | -0.17 (0.616)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.02 (0.784) | -0.09 (0.683)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.16 (0.650) | -0.12 (0.608)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.17 (0.623) | -0.17 (0.595)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.01 (0.749) | -0.05 (0.783)

14. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Score (Temporal Region)
Description: It is evaluated for the temporal region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.29 (0.734) | 1.35 (0.759)
  Day 1 Post-CAE | 1.47 (0.798) | 1.55 (0.850)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.18 (0.601) | 0.21 (0.752)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.12 (0.708) | -0.07 (0.811)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.14 (0.733) | -0.18 (0.806)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.11 (0.714) | -0.23 (0.715)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.03 (0.865) | -0.07 (0.887)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.21 (0.687) | -0.19 (0.827)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.22 (0.659) | -0.29 (0.780)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.03 (0.811) | -0.09 (0.918)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.18 (0.774) | -0.21 (0.817)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.18 (0.774) | -0.23 (0.822)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.00 (0.868) | -0.02 (1.023)

15. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Score (Nasal Region)
Description: It is evaluated for the nasal region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.51 (0.852) | 1.48 (0.823)
  Day 1 Post-CAE | 1.80 (0.903) | 1.82 (0.915)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.29 (0.680) | 0.34 (0.697)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.09 (0.732) | -0.07 (0.655)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.16 (0.772) | -0.16 (0.695)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.14 (0.808) | -0.23 (0.729)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.03 (0.894) | -0.09 (0.830)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.24 (0.801) | -0.22 (0.690)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.28 (0.804) | -0.37 (0.810)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.07 (0.896) | -0.16 (0.905)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.17 (0.751) | -0.16 (0.657)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.20 (0.898) | -0.29 (0.816)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.04 (0.985) | -0.13 (0.862)

16. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining (Corneal Sum)
Description: Corneal sum score is the sum of all regions of the cornea (inferior, superior and central regions). Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 12. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 2.24 (1.711) | 2.33 (1.621)
  Day 1 Post-CAE | 3.22 (2.083) | 3.27 (2.082)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.98 (1.522) | 0.95 (1.433)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.04 (1.663) | -0.16 (1.644)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.32 (1.594) | -0.30 (1.599)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.37 (1.696) | -0.39 (1.846)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.04 (1.875) | -0.08 (1.933)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 306 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.37 (1.513) | -0.47 (1.555)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.44 (1.688) | -0.52 (1.805)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.09 (1.899) | -0.05 (1.884)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.48 (1.502) | -0.51 (1.473)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.55 (1.676) | -0.63 (1.609)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.06 (1.833) | -0.12 (1.900)

17. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining (Conjunctival Sum)
Description: Conjunctival sum score is the sum of all regions of the conjunctiva (temporal and nasal regions). Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 8. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 2.81 (1.428) | 2.83 (1.436)
  Day 1 Post-CAE | 3.28 (1.520) | 3.37 (1.551)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.47 (1.080) | 0.54 (1.181)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.21 (1.235) | -0.15 (1.241)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.30 (1.271) | -0.34 (1.335)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.25 (1.232) | -0.46 (1.142)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.05 (1.442) | -0.16 (1.351)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.44 (1.263) | -0.41 (1.269)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.51 (1.220) | -0.67 (1.261)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.10 (1.409) | -0.25 (1.442)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.35 (1.315) | -0.38 (1.245)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.38 (1.453) | -0.51 (1.383)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.04 (1.581) | -0.14 (1.510)

18. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (All Five Regions: Central, Superior, Inferior, Temporal, Nasal)
Description: Total score was sum of all 5 regions: central, superior, inferior, temporal, and nasal. Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 20. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 5.04 (2.765) | 5.15 (2.643)
  Day 1 Post-CAE | 6.49 (3.166) | 6.64 (3.180)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.45 (2.111) | 1.49 (2.067)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.25 (2.445) | -0.31 (2.468)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.62 (2.435) | -0.63 (2.568)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.62 (2.384) | -0.85 (2.424)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.01 (2.624) | -0.25 (2.593)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 306 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.82 (2.302) | -0.88 (2.376)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.94 (2.389) | -1.19 (2.464)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.19 (2.695) | -0.30 (2.555)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.83 (2.366) | -0.89 (2.217)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.93 (2.586) | -1.15 (2.518)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.11 (2.812) | -0.26 (2.773)

19. Secondary Outcome: Measure Title Change From Baseline in the Ora Calibra® Conjunctival Redness Scale
Description: It is evaluated by the Ora Calibra® conjunctival redness scale for dry eye. The score ranges from 0 to 4 (0=none and 4=severe), where lower score indicates improvement
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 1.53 (0.588) | 1.55 (0.617)
  Day 1 Post-CAE | 1.89 (0.718) | 1.95 (0.739)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.36 (0.511) | 0.40 (0.503)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.13 (0.595) | -0.10 (0.528)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -0.22 (0.650) | -0.18 (0.596)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.37 (0.691) | -0.35 (0.706)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.14 (0.630) | -0.17 (0.578)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.15 (0.609) | -0.16 (0.607)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.31 (0.729) | -0.36 (0.781)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.17 (0.666) | -0.18 (0.620)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 290 | 294
  Change from Baseline: Day 57 (Pre-CAE) | 0.04 (0.565) | -0.05 (0.494)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.07 (0.579) | -0.26 (0.561)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.10 (0.656) | -0.21 (0.677)

20. Secondary Outcome: Change From Baseline in Schirmer's Test
Description: The Schirmer test strip will be placed in the lower temporal lid margin of each eye. Participants will be instructed to close their eyes and After 5 minutes have elapsed, The length of moistened area of schirmer strip will be recorded (mm) for each eye.
Time Frame: Post CAE on baseline (Day 1) and Days 15, 29, and 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Post-CAE | 5.1 (2.80) | 4.9 (2.80)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Post-CAE) | 1.2 (5.41) | 2.0 (5.69)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 305 | 303
  Change from Baseline: Day 29 (Post-CAE) | 2.0 (6.14) | 1.2 (5.26)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 286 | 293
  Change from Baseline: Day 57 (Post-CAE) | 3.2 (7.55) | 2.4 (6.12)

21. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time
Description: Sodium fluorescein solution was instilled into each eye and participants were instructed to blinked several times. The time it takes to form micelles from the time that the eye is opened was noted.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
seconds
  Day 1 Pre-CAE | 2.482 (0.8960) | 2.588 (1.0003)
  Day 1 Post-CAE | 2.444 (0.8056) | 2.504 (0.9018)
  Day 1 (Change from Pre-CAE to Post-CAE) | -0.037 (0.7530) | -0.084 (0.8608)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | 0.175 (1.2459) | 0.190 (1.1859)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | 0.276 (1.4305) | 0.368 (1.3630)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | 0.340 (1.4089) | 0.348 (1.2850)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.058 (1.2997) | -0.021 (1.2701)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | 0.311 (1.3669) | 0.352 (1.5754)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 298 | 293
  Change from Baseline: Day 29 (Post-CAE) | 0.222 (1.1373) | 0.302 (1.2757)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 298 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.125 (1.1118) | -0.071 (1.2797)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 288 | 294
  Change from Baseline: Day 57 (Pre-CAE) | 0.610 (1.3934) | 0.478 (1.2693)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 281 | 289
  Change from Baseline: Day 57 (Post-CAE) | 0.523 (1.1321) | 0.726 (1.6787)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 281 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.085 (1.3655) | 0.246 (1.6429)

22. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI)
Description: The OSDI is a simple 12-question survey that rates the severity of the participant's dry eye disease based on the symptoms. It is assessed on a scale of 0 to 100, with higher score representing greater disability.
Time Frame: Pre-CAE on baseline (Day 1) and Days 15, 29, and 57; Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Day 1 Pre-CAE | 39.7 (19.68) | 39.2 (19.33)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -2.0 (12.50) | -1.5 (12.46)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -2.7 (12.07) | -1.5 (12.81)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -3.7 (13.13) | -2.2 (13.95)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -2.9 (14.69) | -5.3 (13.93)

23. Secondary Outcome: Change From Baseline in Visual Analog Scale (Blurry Vision)
Description: Participants rated ocular symptom of blurry vision by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 37.8 (28.41) | 32.9 (28.67)
  Day 1 Post-CAE | 43.7 (29.37) | 40.5 (29.68)
  Day 1 (Change from Pre-CAE to Post-CAE) | 5.9 (17.70) | 7.6 (18.80)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -2.4 (18.85) | -0.8 (17.90)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -2.8 (20.85) | -1.3 (18.59)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -3.9 (20.70) | -3.1 (18.99)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.9 (23.30) | -2.1 (21.88)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -3.9 (22.40) | -1.3 (20.30)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 293
  Change from Baseline: Day 29 (Post-CAE) | -6.2 (22.30) | -5.2 (21.84)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -2.3 (22.41) | -3.9 (23.19)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -6.5 (22.49) | -5.7 (21.23)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -7.1 (24.39) | -6.3 (24.68)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.3 (22.62) | -0.2 (24.41)

24. Secondary Outcome: Change From Baseline in Visual Analog Scale (Burning/Stinging)
Description: Participants rated ocular symptom of burning/stinging by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 36.6 (28.19) | 35.6 (27.23)
  Day 1 Post-CAE | 49.2 (31.81) | 47.1 (30.02)
  Day 1 (Change from Pre-CAE to Post-CAE) | 12.6 (24.32) | 11.5 (23.00)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -3.7 (18.86) | -3.9 (19.55)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -4.9 (21.12) | -5.7 (19.94)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -5.2 (23.93) | -4.5 (23.80)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.1 (26.13) | 1.5 (24.77)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -6.5 (24.75) | -5.4 (18.45)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 293
  Change from Baseline: Day 29 (Post-CAE) | -5.2 (24.73) | -5.4 (24.50)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 1.5 (29.65) | -0.6 (24.52)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -7.6 (23.03) | -9.1 (21.37)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -6.8 (26.31) | -7.4 (27.83)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 1.1 (28.56) | 1.8 (29.03)

25. Secondary Outcome: Change From Baseline in Visual Analog Scale (Itching)
Description: Participants rated ocular symptom of itching by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 35.9 (27.26) | 35.6 (27.53)
  Day 1 Post-CAE | 42.3 (30.44) | 39.6 (28.83)
  Day 1 (Change from Pre-CAE to Post-CAE) | 6.5 (21.23) | 4.0 (19.81)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -5.1 (20.76) | -4.2 (19.66)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -5.2 (22.62) | -4.6 (21.02)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 307 | 295
  Change from Baseline: Day 15 (Post-CAE) | -7.1 (21.79) | -3.7 (21.96)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 307 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -2.0 (25.24) | 1.0 (23.34)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 307 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -8.4 (22.61) | -5.9 (20.75)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 292
  Change from Baseline: Day 29 (Post-CAE) | -7.8 (24.13) | -5.9 (22.57)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 292
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.5 (26.78) | -0.4 (22.52)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -8.0 (21.70) | -8.3 (23.57)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -8.9 (24.09) | -7.2 (27.69)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.8 (24.68) | 1.3 (26.04)

26. Secondary Outcome: Change From Baseline in Visual Analog Scale (Foreign Body Sensation)
Description: Participants rated ocular symptom of foreign body sensation by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 37.8 (28.96) | 36.6 (28.81)
  Day 1 Post-CAE | 47.5 (30.70) | 42.9 (30.08)
  Day 1 (Change from Pre-CAE to Post-CAE) | 9.7 (21.96) | 6.3 (19.33)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -3.9 (19.98) | -3.6 (21.88)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -5.5 (21.35) | -5.6 (21.37)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -7.9 (24.27) | -2.9 (21.23)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -2.1 (25.53) | 2.5 (23.43)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -6.9 (24.63) | -4.7 (22.85)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 292
  Change from Baseline: Day 29 (Post-CAE) | -9.0 (26.10) | -4.0 (22.44)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 292
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -2.0 (28.75) | 0.6 (22.51)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -7.6 (23.30) | -8.2 (22.70)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -9.1 (25.32) | -5.6 (26.82)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.9 (26.40) | 2.9 (25.60)

27. Secondary Outcome: Change From Baseline in Visual Analog Scale (Eye Dryness)
Description: Participants rated ocular symptom of eye dryness by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 61.4 (24.71) | 59.7 (24.58)
  Day 1 Post-CAE | 74.4 (22.20) | 72.4 (21.45)
  Day 1 (Change from Pre-CAE to Post-CAE) | 13.1 (20.49) | 12.7 (18.58)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -5.5 (19.57) | -3.7 (19.20)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -7.7 (21.44) | -6.8 (19.33)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -5.4 (17.94) | -5.0 (17.45)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 2.5 (23.52) | 1.9 (20.81)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -9.8 (23.24) | -7.4 (22.31)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 293
  Change from Baseline: Day 29 (Post-CAE) | -7.4 (20.28) | -6.9 (19.91)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 2.6 (25.92) | 0.6 (21.09)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -12.9 (24.74) | -11.3 (23.01)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -10.6 (22.58) | -10.3 (24.63)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 2.3 (25.84) | 1.2 (24.96)

28. Secondary Outcome: Change From Baseline in Visual Analog Scale (Photophobia)
Description: Participants rated ocular symptom of photophobia by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 40.4 (30.20) | 37.8 (30.73)
  Day 1 Post-CAE | 46.0 (31.33) | 43.5 (30.48)
  Day 1 (Change from Pre-CAE to Post-CAE) | 5.6 (19.67) | 5.7 (17.70)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -3.2 (16.91) | -3.6 (17.03)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -3.4 (18.66) | -3.6 (18.58)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -4.0 (21.77) | -4.9 (22.13)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.4 (22.09) | -1.3 (20.38)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -6.3 (20.75) | -4.9 (21.05)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 293
  Change from Baseline: Day 29 (Post-CAE) | -6.5 (21.85) | -7.0 (23.42)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.0 (22.25) | -2.1 (22.44)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -7.4 (21.60) | -7.6 (20.66)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -8.2 (22.51) | -9.5 (23.72)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.4 (22.72) | -1.9 (22.26)

29. Secondary Outcome: Change From Baseline in Visual Analog Scale (Pain)
Description: Participants rated ocular symptom of pain by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 27.7 (26.43) | 26.2 (25.34)
  Day 1 Post-CAE | 39.3 (31.31) | 37.0 (29.17)
  Day 1 (Change from Pre-CAE to Post-CAE) | 11.6 (22.26) | 10.8 (21.13)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 312
  Change from Baseline: Day 8 | -3.7 (17.44) | -2.9 (19.27)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 305
  Change from Baseline: Day 15 (Pre-CAE) | -3.5 (20.36) | -4.0 (19.52)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -5.2 (23.17) | -5.8 (21.95)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 295
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -1.3 (24.59) | -1.9 (21.55)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -5.7 (22.52) | -5.4 (20.52)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 297 | 293
  Change from Baseline: Day 29 (Post-CAE) | -6.3 (22.39) | -9.0 (23.24)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 297 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.6 (24.88) | -3.6 (23.73)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 293 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -5.3 (21.66) | -7.3 (22.61)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 280 | 289
  Change from Baseline: Day 57 (Post-CAE) | -7.7 (25.24) | -8.3 (25.19)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 280 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -1.8 (25.64) | -0.8 (26.50)

30. Secondary Outcome: Change From Baseline in Ocular Discomfort Scale
Description: It was assessed by the Ora Calibra® ocular discomfort scale. The score ranges from 0 to 4 (0=none and 4=severe), where lower score indicates improvement.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 2.6 (0.98) | 2.5 (1.06)
  Day 1 Post-CAE | 3.6 (0.59) | 3.6 (0.64)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.0 (1.07) | 1.1 (1.12)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.3 (1.20) | -0.2 (1.11)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.5 (1.18) | -0.3 (1.18)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 294
  Change from Baseline: Day 15 (Post-CAE) | -0.2 (0.77) | -0.1 (0.74)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 293
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.3 (1.32) | 0.1 (1.36)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.4 (1.30) | -0.2 (1.23)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 294
  Change from Baseline: Day 29 (Post-CAE) | -0.2 (0.73) | -0.2 (0.84)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 294
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.2 (1.44) | 0.0 (1.38)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.5 (1.29) | -0.5 (1.24)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 279 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.4 (0.91) | -0.3 (0.95)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 279 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.41) | 0.2 (1.37)

31. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Overall Ocular Discomfort)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. At each day during the at-home dosing period, subjects will grade the severity of their dry eye syndrome symptoms in the morning and in the evening, before instilling the study drug. Participants rated the severity of overall ocular discomfort on 0 to 5 scale, where 0=none and 5=severe.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 2.8 (0.94) | 2.8 (1.00)
  Day 1 Post-CAE | 3.7 (0.82) | 3.7 (0.79)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.9 (0.98) | 0.9 (0.98)
  Change from Baseline: Day 8: number analyzed (Participants) | 313 | 314
  Change from Baseline: Day 8 | -0.2 (1.05) | -0.2 (1.03)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.4 (1.09) | -0.3 (0.99)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.2 (0.95) | -0.3 (0.82)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 294
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.2 (1.35) | 0.1 (1.17)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.4 (1.14) | -0.3 (1.20)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (0.86) | -0.3 (0.89)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.1 (1.29) | 0.0 (1.40)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.4 (1.21) | -0.5 (1.14)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 279 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.4 (1.01) | -0.4 (1.04)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 279 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.31) | 0.1 (1.21)

32. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Burning)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. At each day during the at-home dosing period, subjects graded the severity of their dry eye syndrome symptoms in the morning and in the evening, before instilling the study drug. Participants rated the severity of burning on 0 to 5 scale, where 0=none and 5=severe.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 1.7 (1.43) | 1.7 (1.38)
  Day 1 Post-CAE | 2.6 (1.56) | 2.6 (1.56)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.9 (1.34) | 0.9 (1.22)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.1 (1.14) | -0.2 (1.08)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.2 (1.18) | -0.2 (1.15)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.3 (1.18) | -0.3 (1.20)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 294
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.1 (1.50) | -0.1 (1.43)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.3 (1.18) | -0.2 (1.16)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (1.26) | -0.3 (1.25)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.1 (1.57) | -0.2 (1.55)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.3 (1.19) | -0.4 (1.25)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 279 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.3 (1.37) | -0.4 (1.36)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 279 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.0 (1.49) | 0.0 (1.61)

33. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Dryness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. At each day during the at-home dosing period, subjects graded the severity of their dry eye syndrome symptoms in the morning and in the evening, before instilling the study drug. Participants rated the severity of dryness on 0 to 5 scale, where 0=none and 5=severe.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 3.2 (1.05) | 3.2 (0.97)
  Day 1 Post-CAE | 3.9 (0.89) | 3.9 (0.88)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.8 (0.97) | 0.8 (0.95)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.2 (0.98) | -0.3 (1.05)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.4 (1.01) | -0.4 (0.99)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.2 (0.85) | -0.2 (0.78)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 294
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.1 (1.20) | 0.1 (1.11)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.4 (1.16) | -0.4 (1.22)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.2 (0.91) | -0.3 (0.92)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.2 (1.22) | 0.1 (1.38)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.5 (1.22) | -0.6 (1.18)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 279 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.4 (1.12) | -0.5 (1.10)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 279 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.34) | 0.1 (1.34)

34. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Grittiness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. At each day during the at-home dosing period, subjects graded the severity of their dry eye syndrome symptoms in the morning and in the evening, before instilling the study drug. Participants rated the severity of grittiness on 0 to 5 scale, where 0=none and 5=severe.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 2.1 (1.42) | 2.1 (1.43)
  Day 1 Post-CAE | 2.7 (1.49) | 2.6 (1.55)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.6 (1.14) | 0.5 (1.16)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.3 (1.05) | -0.2 (1.17)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.3 (1.12) | -0.3 (1.07)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.3 (1.20) | -0.2 (1.06)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 294
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.0 (1.43) | 0.1 (1.31)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.4 (1.14) | -0.3 (1.15)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (1.20) | -0.3 (1.19)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.1 (1.40) | 0.0 (1.37)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.4 (1.15) | -0.4 (1.20)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 279 | 289
  Change from Baseline: Day 57 (Post-CAE) | -0.4 (1.29) | -0.3 (1.32)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 279 | 289
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.37) | 0.1 (1.46)

35. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Stinging)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. At each day during the at-home dosing period, subjects graded the severity of their dry eye syndrome symptoms in the morning and in the evening, before instilling the study drug. Participants rated the severity of stinging on 0 to 5 scale, where 0=none and 5=severe.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
mm
  Day 1 Pre-CAE | 1.6 (1.42) | 1.6 (1.32)
  Day 1 Post-CAE | 2.3 (1.55) | 2.4 (1.52)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.8 (1.10) | 0.8 (1.11)
  Change from Baseline: Day 8: number analyzed (Participants) | 314 | 314
  Change from Baseline: Day 8 | -0.1 (1.00) | -0.1 (1.03)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 313 | 304
  Change from Baseline: Day 15 (Pre-CAE) | -0.2 (1.07) | -0.3 (1.01)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 308 | 295
  Change from Baseline: Day 15 (Post-CAE) | -0.3 (1.15) | -0.3 (1.17)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 308 | 294
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.1 (1.41) | 0.0 (1.32)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 308 | 304
  Change from Baseline: Day 29 (Pre-CAE) | -0.3 (1.16) | -0.3 (1.05)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 296 | 293
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (1.30) | -0.5 (1.26)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 296 | 293
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.0 (1.48) | -0.2 (1.38)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 295 | 294
  Change from Baseline: Day 57 (Pre-CAE) | -0.4 (1.23) | -0.4 (1.09)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 277 | 288
  Change from Baseline: Day 57 (Post-CAE) | -0.3 (1.24) | -0.5 (1.31)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 277 | 288
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.38) | 0.0 (1.43)

36. Secondary Outcome: Ora Calibra® Drop Comfort Scale
Description: Ora Calibra® drop comfort scale ranges from 0 to 10. A score of 0 indicates comfortable and 10 indicates uncomfortable. Lower score indicated better comfort level.
Time Frame: Upon instillation and 1 and 2 minutes post-instillation on Day 1
Population: The ITT Population with available data. The analysis was carried out with observed data only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 318 | 319
score on a scale
  Upon instillation on Day 1 | 3.5 (2.75) | 3.5 (2.79)
  1 minute post-instillation on Day 1 | 2.5 (2.32) | 2.5 (2.12)
  2 minutes post-instillation on Day 1 | 2.1 (2.19) | 2.0 (2.02)

37. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Overall Ocular Discomfort)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of overall ocular discomfort twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Day -14 to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 310 | 311
score on a scale
  Day -14 - Day -1 (Baseline) Daily Average | 2.7 (0.96) | 2.7 (1.02)
  Day 1 - Day 7, Daily Average Change from Baseline: number analyzed (Participants) | 309 | 307
  Day 1 - Day 7, Daily Average Change from Baseline | -0.1 (0.49) | -0.1 (0.52)
  Day 8 - Day 14, Daily Average Change from Baseline: number analyzed (Participants) | 307 | 308
  Day 8 - Day 14, Daily Average Change from Baseline | -0.2 (0.56) | -0.1 (0.58)
  Day 15 - Day 21, Daily Average Change from Baseline: number analyzed (Participants) | 305 | 304
  Day 15 - Day 21, Daily Average Change from Baseline | -0.2 (0.66) | -0.2 (0.70)
  Day 22 - Day 28, Daily Average Change from Baseline: number analyzed (Participants) | 304 | 298
  Day 22 - Day 28, Daily Average Change from Baseline | -0.3 (0.71) | -0.3 (0.79)
  Day 29 - Day 35, Daily Average Change from Baseline: number analyzed (Participants) | 301 | 297
  Day 29 - Day 35, Daily Average Change from Baseline | -0.3 (0.76) | -0.2 (0.80)
  Day 36 - Day 42, Daily Average Change from Baseline: number analyzed (Participants) | 288 | 293
  Day 36 - Day 42, Daily Average Change from Baseline | -0.3 (0.77) | -0.3 (0.85)
  Day 43 - Day 49, Daily Average Change from Baseline: number analyzed (Participants) | 284 | 290
  Day 43 - Day 49, Daily Average Change from Baseline | -0.3 (0.83) | -0.4 (0.89)
  Day 50 - Day 56, Daily Average Change from Baseline: number analyzed (Participants) | 282 | 289
  Day 50 - Day 56, Daily Average Change from Baseline | -0.3 (0.83) | -0.4 (0.93)

38. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Burning)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of burning twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Day -14 to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 316 | 318
score on a scale
  Day -14 - Day -1 (Baseline) Daily Average | 1.9 (1.21) | 1.8 (1.21)
  Day 1 - Day 7, Daily Average Change from Baseline: number analyzed (Participants) | 315 | 317
  Day 1 - Day 7, Daily Average Change from Baseline | -0.1 (0.44) | -0.1 (0.53)
  Day 8 - Day 14, Daily Average Change from Baseline: number analyzed (Participants) | 313 | 316
  Day 8 - Day 14, Daily Average Change from Baseline | -0.2 (0.58) | -0.2 (0.60)
  Day 15 - Day 21, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 310
  Day 15 - Day 21, Daily Average Change from Baseline | -0.2 (0.63) | -0.2 (0.69)
  Day 22 - Day 28, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 304
  Day 22 - Day 28, Daily Average Change from Baseline | -0.3 (0.69) | -0.3 (0.75)
  Day 29 - Day 35, Daily Average Change from Baseline: number analyzed (Participants) | 308 | 302
  Day 29 - Day 35, Daily Average Change from Baseline | -0.3 (0.71) | -0.3 (0.80)
  Day 36 - Day 42, Daily Average Change from Baseline: number analyzed (Participants) | 297 | 299
  Day 36 - Day 42, Daily Average Change from Baseline | -0.3 (0.73) | -0.3 (0.83)
  Day 43 - Day 49, Daily Average Change from Baseline: number analyzed (Participants) | 293 | 296
  Day 43 - Day 49, Daily Average Change from Baseline | -0.3 (0.78) | -0.3 (0.87)
  Day 50 - Day 56, Daily Average Change from Baseline: number analyzed (Participants) | 289 | 294
  Day 50 - Day 56, Daily Average Change from Baseline | -0.3 (0.82) | -0.4 (0.92)

39. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Dryness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of dryness twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Day -14 to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 316 | 318
score on a scale
  Day -14 - Day -1 (Baseline) Daily Average | 3.0 (0.94) | 2.9 (0.97)
  Day 1 - Day 7, Daily Average Change from Baseline: number analyzed (Participants) | 315 | 317
  Day 1 - Day 7, Daily Average Change from Baseline | -0.1 (0.47) | -0.1 (0.46)
  Day 8 - Day 14, Daily Average Change from Baseline: number analyzed (Participants) | 313 | 316
  Day 8 - Day 14, Daily Average Change from Baseline | -0.3 (0.58) | -0.2 (0.57)
  Day 15 - Day 21, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 310
  Day 15 - Day 21, Daily Average Change from Baseline | -0.3 (0.66) | -0.3 (0.68)
  Day 22 - Day 28, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 304
  Day 22 - Day 28, Daily Average Change from Baseline | -0.4 (0.74) | -0.4 (0.74)
  Day 29 - Day 35, Daily Average Change from Baseline: number analyzed (Participants) | 308 | 302
  Day 29 - Day 35, Daily Average Change from Baseline | -0.4 (0.78) | -0.3 (0.77)
  Day 36 - Day 42, Daily Average Change from Baseline: number analyzed (Participants) | 297 | 299
  Day 36 - Day 42, Daily Average Change from Baseline | -0.5 (0.81) | -0.4 (0.84)
  Day 43 - Day 49, Daily Average Change from Baseline: number analyzed (Participants) | 293 | 296
  Day 43 - Day 49, Daily Average Change from Baseline | -0.5 (0.88) | -0.5 (0.88)
  Day 50 - Day 56, Daily Average Change from Baseline: number analyzed (Participants) | 289 | 294
  Day 50 - Day 56, Daily Average Change from Baseline | -0.5 (0.88) | -0.5 (0.93)

40. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Grittiness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of grittiness twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Day -14 to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 316 | 318
score on a scale
  Day -14 - Day -1 (Baseline) Daily Average | 2.1 (1.26) | 2.0 (1.27)
  Day 1 - Day 7, Daily Average Change from Baseline: number analyzed (Participants) | 315 | 317
  Day 1 - Day 7, Daily Average Change from Baseline | -0.2 (0.49) | -0.1 (0.57)
  Day 8 - Day 14, Daily Average Change from Baseline: number analyzed (Participants) | 313 | 316
  Day 8 - Day 14, Daily Average Change from Baseline | -0.3 (0.64) | -0.2 (0.64)
  Day 15 - Day 21, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 310
  Day 15 - Day 21, Daily Average Change from Baseline | -0.3 (0.69) | -0.2 (0.71)
  Day 22 - Day 28, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 304
  Day 22 - Day 28, Daily Average Change from Baseline | -0.4 (0.75) | -0.3 (0.77)
  Day 29 - Day 35, Daily Average Change from Baseline: number analyzed (Participants) | 308 | 302
  Day 29 - Day 35, Daily Average Change from Baseline | -0.4 (0.77) | -0.3 (0.79)
  Day 36 - Day 42, Daily Average Change from Baseline: number analyzed (Participants) | 297 | 299
  Day 36 - Day 42, Daily Average Change from Baseline | -0.4 (0.76) | -0.3 (0.85)
  Day 43 - Day 49, Daily Average Change from Baseline: number analyzed (Participants) | 293 | 296
  Day 43 - Day 49, Daily Average Change from Baseline | -0.4 (0.84) | -0.4 (0.88)
  Day 50 - Day 56, Daily Average Change from Baseline: number analyzed (Participants) | 289 | 294
  Day 50 - Day 56, Daily Average Change from Baseline | -0.4 (0.85) | -0.4 (0.93)

41. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Stinging)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of stinging twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Day -14 to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 316 | 318
score on a scale
  Day -14 - Day -1 (Baseline) Daily Average | 1.7 (1.25) | 1.7 (1.23)
  Day 1 - Day 7, Daily Average Change from Baseline: number analyzed (Participants) | 315 | 317
  Day 1 - Day 7, Daily Average Change from Baseline | -0.1 (0.48) | -0.1 (0.53)
  Day 8 - Day 14, Daily Average Change from Baseline: number analyzed (Participants) | 313 | 316
  Day 8 - Day 14, Daily Average Change from Baseline | -0.3 (0.62) | -0.2 (0.60)
  Day 15 - Day 21, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 310
  Day 15 - Day 21, Daily Average Change from Baseline | -0.3 (0.68) | -0.3 (0.65)
  Day 22 - Day 28, Daily Average Change from Baseline: number analyzed (Participants) | 311 | 304
  Day 22 - Day 28, Daily Average Change from Baseline | -0.4 (0.72) | -0.3 (0.70)
  Day 29 - Day 35, Daily Average Change from Baseline: number analyzed (Participants) | 308 | 302
  Day 29 - Day 35, Daily Average Change from Baseline | -0.4 (0.74) | -0.3 (0.73)
  Day 36 - Day 42, Daily Average Change from Baseline: number analyzed (Participants) | 297 | 299
  Day 36 - Day 42, Daily Average Change from Baseline | -0.4 (0.76) | -0.3 (0.79)
  Day 43 - Day 49, Daily Average Change from Baseline: number analyzed (Participants) | 293 | 296
  Day 43 - Day 49, Daily Average Change from Baseline | -0.4 (0.79) | -0.4 (0.82)
  Day 50 - Day 56, Daily Average Change from Baseline: number analyzed (Participants) | 289 | 294
  Day 50 - Day 56, Daily Average Change from Baseline | -0.4 (0.84) | -0.4 (0.86)

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks
Arm/Group | 0.25% HL036 Ophthalmic Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 1/318 | 0/319
Serious Adverse Events (participants affected / at risk) | 5/318 | 4/319
Other Adverse Events (participants affected / at risk) | 78/318 | 76/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25% HL036 Ophthalmic Solution (N=318) | Placebo (N=319)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25% HL036 Ophthalmic Solution (N=318) | Placebo (N=319)
Instillation site pain (General disorders) | 62 | 58
Visual acuity reduced (Eye disorders) | 16 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT03846453/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03846453/SAP_001.pdf